CLINICAL TRIAL: NCT04787172
Title: Role of the Multi-Slice Computed Tomography in Evaluation of the Congenital Cardiovascular Anomalies
Brief Title: Role of the MSCT in Evaluation of the Congenital Cardiovascular Anomalies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ali Gamal, specialist, Assiut University
Other Study IDs: MSCT in congenital CVA
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: MSCT in Congenital Cardiovascular Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Multi Slice computed tomography — use of MSCT as a diagnostic tool in evaluation of patients with congenital cardiovascular anomalies

SUMMARY:
Congenital heart diseases (CHDs) are considered as the most common congenital birth defects, comprising 1% of all live births . Echocardiography remains a first-line non-invasive imaging tool for establishing the diagnosis and follow-up in most patients .This method is operator dependent and limited by an acoustic window .

Traditional angiography is typically utilized as the gold standard modality for diagnosing CHD, but it is an invasive method and need general anseathsia with dose of radiation exposure .After recent developments in CT and MR technologies, cardiac catheterization is no longer necessary for diagnosis .

DETAILED DESCRIPTION:
The interpretation of cardiovascular structures on cardiac CT scan studies is similar to that for echocardiography, however, it is not limited by the acoustic window or operator dependent like ultrasonography. In addition to the anatomic information, a cardiac CT scan provides hemodynamic information, including extracardiac and intra-cardiac shunts. It also enables the systematic evaluation of other thoracic structures like cardiovascular structures, the airways and the lungs by using maximum and minimum intensity projections to delineate the vascular and airway structures, respectively. Extra-cardiac great vessels can be evaluated along their length; thus augmenting the role of cardiac CT scans in children with congenital heart diseases .Inspite of the poorer temporal resolution of cardiac CTA compared to echocardiography, yet the combination of rapid acquisition time, increased anatomic coverage, high spatial resolution, multiplanar reformation and 3D capability combined with a flexible ECG synchronization have improved the image quality of cardiac CT scans and minimizing the patient risks. Multidetector computed tomography has greatly advanced the noninvasive diagnosis of these anomalies in pediatric patient, thus makes MDCT an ideal non- invasive method for evaluating pediatric patients .

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from congenital cardiovascular diseases diagnosed either clinically or by echocardiographic examination.

Exclusion Criteria:

* orthopenic patient patients with hypersensitivity to contrast , medium and poor renal function .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending to the cardiovascular departement and diagnosed as congenital cardiovascular anomalies
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of the MSCT in congenital cardiovascular anomalies | baseline
  comparison between sensitivity and accuracy of MSCT in detection of congenital cardiovascular anomalies with detection rate by cardiac catheterization or surgery

REFERENCES:
- [Result] Goitein O, Salem Y, Jacobson J, Goitein D, Mishali D, Hamdan A, Kuperstein R, Di Segni E, Konen E. The role of cardiac computed tomography in infants with congenital heart disease. Isr Med Assoc J. 2014 Mar;16(3):147-52. PMID 24761701